CLINICAL TRIAL: NCT03497832
Title: Diurnal Variations of Cerebral Metabolite Concentrations in Proton Magnetic Resonance Spectroscopy
Brief Title: Diurnal Variations of Brain Metabolite Concentrations in 1H-MRS
Acronym: Dyn24
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-A02804-49
Record Dates: First submitted 2018-03-09; First posted 2018-04-13 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Diurnal Variations of Cerebral Metabolite
Keywords: Proton Magnetic Resonance Spectroscopy
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: magnetic resonance spectroscopy (MRI) — Each healthy subject will get 3 MRI examinations at 7:30, 13:30 and 18:00. Each MRI scan lasts an average of 20 minutes.

SUMMARY:
Proton Magnetic Resonance Spectroscopy (1H-MRS) is a magnetic resonance imaging (MRI) technique. It allows the quantification of cerebral metabolite concentrations. Currently, MRS-1H is used regardless of the examination schedule. However, it is not possible to say if the brain metabolite concentrations are stable over 24 hours. Thus, the main objective was to study the diurnal variation of cerebral metabolite concentrations in 1H-MRS in healthy subjects.

Moreover, the investigators also want to investigate the association between choline concentrations (Cho, parameter reflecting membrane metabolism) in 1H-MRS and fractional anisotropy (AF) values, obtained with the diffusion tensor imaging sequence (DTI), in the white matter of the centrum ovale. The results obtained from this objective will allow to obtain reference values of an estimate of the association between Cho concentrations and AF values in healthy subjects. These data are intended to improve the diagnostic and therapeutic management of patients with neurological pathologies.

DETAILED DESCRIPTION:
Currently, it is not possible to say if the brain metabolite concentrations are stable over 24 hours in 1H-MRS. Few studies, with small samples (< 10 subjects), have investigated this point. Their conclusions remain inconsistent. Without an available study with sufficient statistical power, it is not currently possible to state that concentrations of brain metabolites are stable over 24 hours. Therefore, it is not possible to formally conclude on differences in concentrations of metabolites between a healthy subject and a patient.

It is known that the human circadian rhythm leads to changes on many parameters such as hormonal secretions (TSH, cortisol, melatonin, growth hormone, and carbohydrate metabolism) and body temperature. It therefore seemed relevant to choose 3 of the most critical periods of the human circadian rhythm (7:30, 13:30 and 18:00) to assess the diurnal variations of cerebral metabolite in 1H-MRS. The DTI sequence will only be performed once.

The study will take place at the University Hospital of Poitiers, in the department of Medical Imaging. 3 appointments are planned: the pre-inclusion one D0, the inclusion one D1 including the signature of the consent, and the D3 one for the realization of the 3 MRIs at 7:30 am, 1:30 pm and 6 pm. Each MRI scan lasts an average of 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-45 years
* Voluntary subjects, without guardianship or curatorship or subordination
* Subjects benefiting from a Social Security scheme or benefiting from it through a relative
* Informed and signed consent by the subject after a clear and fair information of the study

Exclusion Criteria:

* Age < 25 years or > 45 years
* Current participation in another clinical research study
* Subjects not benefiting from a Social Security scheme or not benefiting from it through a relative
* Subjects benefiting from enhanced protection, namely minors, pregnant women, nursing mothers, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social institution, adults under legal protection, and patients in emergencies.
* Pregnant or nursing women, women of childbearing age who do not have effective contraception (hormonal / mechanical: oral, injectable, transcutaneous, implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, total ovariectomy )
* Neurological, psychiatric, endocrinological, cardiac, pulmonary disorders.
* Unbalanced sleep disorders: untreated obstructive sleep apnea, insomnia, major delayed or advanced sleep phase, shift work with irregular rhythms.
* Taking any type of treatment, except oral contraception for women.
* Any contraindication to performing an MRI examination: pregnancy, ocular metallic foreign body (accidental blisters or others); Tattooing for a part of the face or skull, pacemaker (cardiac simulator), neurostimulator, cochlear implants and in general any implanted medical equipment; metallic cardiac valve, vascular clips formerly implanted on cranial aneurysm.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Description of diurnal variations of brain metabolite concentrations in 1H-MRS | 1 day
  The primary outcome is to describe the diurnal variation of N-acetylaspartate (NAA), choline (Cho), creatine (Cr), gamma-aminobutyric acid (GABA) and glutamate at 7:30 am, 1:30 pm and 6 pm, in the basal ganglia, the anterior and posterior cingulate cortex, the insular cortex, the white matter in healthy subjects. The data will be collected at D3.

SECONDARY OUTCOMES:
investigation of the association between Cho concentrations and AF values in the white matter of the centrum ovale. | 1 day
  investigation of the association between Cho concentrations and AF values in the white matter of the centrum ovale.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Poitiers, France